CLINICAL TRIAL: NCT07246252
Title: Phase I Comparison of Pharmacokinetics, Safety, and Immunogenicity of Process-Changed CMAB007 and Xolair in a Randomized, Double-blind, Parallel Controlled, Single-dose Study in Healthy Chinese Male Subjects
Brief Title: Compare the PK, Safety, and Immunogenicity of Process-Changed CMAB007 and Xolair in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taizhou Mabtech Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMAB007-004
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers (HV)
MeSH Terms: interventions — Omalizumab

STUDY DESIGN:
Intervention Model Description: Biological: Process-Changed CMAB007 Biological: Xolair
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Process-Changed CMAB007 (Experimental): 150 mg Subcutaneous injection
  Interventions: Biological: Process-Changed CMAB007
- Xolair (Active Comparator): 150 mg Subcutaneous injection
  Interventions: Biological: Xolair (omalizumab)

INTERVENTIONS:
Biological: Process-Changed CMAB007 — for subcutaneous injection only
  Arms: Process-Changed CMAB007
Biological: Xolair (omalizumab) — for subcutaneous injection only
  Arms: Xolair

SUMMARY:
A phase 1, randomized, double-blind, parallel group, single-dose study to compare the pharmacokinetics, safety and immunogenicity of two formulations of Omalizumab (Process-Changed CMAB007 and Xolair) in healthy subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-controlled, single-dose phase I clinical study in healthy Chinese male subjects. A total of 114 subjects were planned to be enrolled and randomly assigned to the test group or the control group in a 1:1 ratio. Subjects in both groups received a single subcutaneous injection of Process-Changed CMAB007 or Xolair(Omalizumab) 150 mg, respectively. Subjects in both groups were observed for 106 days after administration to evaluate similarities in PK, safety, and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, age ranged 18 to 45 years (both inclusive) when sign the informed consent form.
2. Subjects with body weight of ≥50 kg and ≤ 75 kg and BMI ≥20.0 and ≤ 26.0 kg/m2 (both inclusive).
3. Subjects have the ability to understand the full characteristics and objectives of the study, including the possible risks and side effects of the study; moreover, subjects can communicate well with researchers and complete the research according to the regulations.
4. Subjects must be informed consent of the study and voluntarily sign informed consent form (name and time) prior to the study.

Exclusion Criteria:

1. After medical examination (vital signs, physical examination, electrocardiogram, positive chest X-radiography, abdominal B-ultrasound, and various laboratory examinations including blood routine, urine routine, blood biochemistry and total IgE, etc.), any examination item was judged abnormal by the investigator and had clinical significance.
2. Subjects with a history of clinically significant drug or food allergies, a history of specific allergic diseases (e.g., asthma, urticaria, eczematous dermatitis), allergic rhinitis, or a known allergy to any component of the investigational drug or latex (the syringe needle cover contains latex) as determined by the investigator..
3. Those who have a history of serious diseases including but not limited to cardiovascular system, respiratory system, digestive system, urogenital system, endocrine system, immune system, mental or nervous system (eg, epilepsy, etc), or currently have any of the above diseases or active infected diseases, or any other disease or medical condition that may interfere with the results of the trial, such as hereditary bleeding tendency, coagulation disorders or history of blood clots or bleeding.
4. History of malignant neoplasms within the last 5 years (other than completely resected basal cell or squamous cell carcinoma of the skin in situ).
5. Any one of HBV surface antigen, HIV antibody, HCV antibody and treponema pallidum antibody is positive.
6. Anti-nuclear antibody is positive.
7. Fecal parasite test is positive.
8. Those who smoke more than 10 cigarettes per day on average in the 6 months before screening.
9. Alcoholics or regular drinkers within 3 months before the test, i.e. those who drink more than 14 unites of alcohol per week (14 bottles of 360 ml beer or 45 ml spirits with 40% alcohol or 150 ml wine), or whose alcohol breath test is positive.
10. Drug abusers, or use of soft drugs within 3 months prior to screening or hard drugs within 1 year prior the trial, or excessive daily consumption of tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup =250mL) in the 3 months prior to screening, or positive urine drug screening.
11. Surgery within 4 weeks prior to screening; Or plan to have surgery during the study period.
12. Use of any prescription drug, over-the-counter drug or health product or vaccine within 4 weeks prior to screening, or who plan to receive live vaccine during the study period, or prior use of drug within 5 half-lives, whichever is longer.
13. Subjects who have donated blood (including whole blood or component blood) or experienced blood loss of more than 400 mL within 3 months prior to screening, or have received a blood transfusion; or who have donated blood (including component blood) or experienced blood loss of more than 200 mL within 1 month prior to screening; or who plan to donate blood during the study period..
14. Those who have been enrolled in other clinical studies or less than 3 months since the end of the most recent clinical study.
15. Subjects and their partners were not willing to use medically approved contraceptive methods within 6 months of study administration, or partners plan to become pregnant, or subjects plan to donate sperm.
16. Use of anti-IgE mab within 12 months, or any biological agent within 3 months prior to screening.
17. The investigator judges the subject inappropriate to be included in this study or other reasons not eligible to complete the study.
18. Employees or related personnel of the research unit, sponsor or contract research organization.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Zero (0) Hours Extrapolated to infinite time | up to 2520 hours
  Area Under the Plasma Concentration-time Curve From Zero (0) Hours Extrapolated to infinite time After the Single injection of Omalizumab
Maximum Concentration of Omalizumab | up to 2520 hours
  Maximum Concentration After the Single Injection of Omalizumab

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Zero (0) Hours to 2520 Hours | up to 2520 hours
  Area Under the Plasma Concentration-time Curve From Zero (0) Hours to 2520 Hours After the Single Injection of Omalizumab
Time to Maximum Concentration of Omalizumab | up to 2520 hours
  Time to Maximum Concentration of Omalizumab after the Single Injection of Omalizumab
Half time | up to 2520 hours
  Half-time after the Single Injection of Omalizumab
Terminal elimination rate constant (λz) | up to 2520 hours
  Terminal elimination rate constant (λz) after the Single Injection of Omalizumab
Apparent total body clearance (CL/F) | up to 2520 hours
  Apparent total body clearance (CL/F) after the Single Injection of Omalizumab
Apparent total distribution (Vd/F) | up to 2520 hours
  Apparent total distribution (Vd/F) after the Single Injection of Omalizumab
anti-drug antibodies (ADA) | up to 2520 hours
  ADA Positive Rate after the Single Injection of Omalizumab
Neutralization antibodies (Nab) | up to 2520 hours
  Neutralizing Antibody Positive Rate after the Single Injection of Omalizumab
Percentage and Severity of Participants with Adverse Events | up to 2520 hours
  Total Frequency and Severity of Adverse Events/Serious Adverse Events Within the Whole Time of the Study

CONTACTS AND LOCATIONS:
Overall Officials: Jingying Jia, Ph.D, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai, China

IPD SHARING:
Plan to Share IPD: No